CLINICAL TRIAL: NCT01081145
Title: A Phase 3, Double-blind, Placebo-controlled, Multicentre, Randomised Withdrawal, Long-term Maintenance of Efficacy and Safety Study of Extended-release Guanfacine Hydrochloride in Children and Adolescents Aged 6-17 With Attention Deficit/Hyperactivity Disorder
Brief Title: Maintenance of Efficacy of Extended-Release Guanfacine HCl in Children and Adolescents With Attention-deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPD503-315; 2009-018161-12 (EudraCT Number)
Record Dates: First submitted 2010-03-03; First posted 2010-03-05 (Estimated); Results first posted 2014-06-09 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Attention-deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Extended-release Guanfacine HCl (Experimental)
  Interventions: Drug: Extended-release Guanfacine Hydrochloride
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Extended-release Guanfacine Hydrochloride — The test product will be provided as 1, 2, 3, and 4mg tablets. Subjects will be administered a once-daily dose between 1-7mg/day depending on age and weight.
  Arms: Extended-release Guanfacine HCl
Other: Placebo — Matching placebo will be provided as 1, 2, 3, and 4mg tablets. Subjects will be administered a once-daily dose of placebo between 1-7mg/day depending on age and weight.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the long-term maintenance of efficacy of Extended-Release Guanfacine HCl in children and adolescents (6-17 years) with attention-deficit/hyperactivity disorder (ADHD) who respond to an initial open-label, short term treatment with SPD503.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 6-17 years at the time of consent/assent at Screening/Visit 1.
2. Subject's parent or legally authorised representative (LAR) must provide signature of informed consent, and there must be documentation of assent (if applicable) by the subject indicating that the subject is aware of the investigational nature of the study and the required procedures and restrictions, in accordance with the International Conference on Harmonisation (ICH) Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations before completing any study-related procedures at Screening/Visit 1.
3. Subject meets DSM-IV-TR criteria for a primary diagnosis of ADHD, combined subtype, hyperactive/impulsive subtype, or inattentive sub-type based on a detailed psychiatric evaluation using the Kiddie Schedule for Affective Disorders and Schizophrenia-Present and Lifetime version (K-SADS-PL).
4. Subject has a minimum ADHD-RS-IV total score of 32 at Enrolment/Visit 2.
5. Subject has a minimum CGI-S score of 4 at Enrolment/Visit 2.
6. Subject is functioning at an age-appropriate level intellectually, as deemed by the Investigator.
7. Subject and parent/LAR understand, are willing, able, and likely to fully comply with the study requirements, procedures, and restrictions defined in this protocol.
8. Subject is able to swallow intact tablets.
9. Subject who is a female of child-bearing potential (FOCP), defined as 9 years of age or <9 years of age and is post-menarchal, must have a negative serum beta Human Chorionic Gonadotropin (hCG) pregnancy test at Screening/Visit 1 and a negative urine pregnancy test at Enrolment/Visit 2 and agree to comply with any applicable contraceptive requirements of the protocol.
10. Subject has a supine and standing BP measurement within the 95th percentile for age, gender, and height.

Exclusion Criteria:

1. Subject has a current, controlled (requiring a prohibited medication or behavioural modification program) or uncontrolled, comorbid psychiatric diagnosis, except oppositional defiant disorder (ODD), including any severe comorbid Axis II disorders or severe Axis I disorders such as post traumatic stress disorder, bipolar illness, psychosis, pervasive developmental disorder, obsessive-compulsive disorder, substance abuse disorder, or other symptomatic manifestations or lifetime history of bipolar illness, psychosis, or conduct disorder that, in the opinion of the Investigator, contraindicate SPD503 treatment or confound efficacy or safety assessments.
2. Subject has any condition or illness including clinically significant abnormal Screening/Visit 1 laboratory values which, in the opinion of the Investigator, represents an inappropriate risk to the subject and/or could confound the interpretation of the study.
3. Subject has a known history or presence of structural cardiac abnormalities, serious heart rhythm abnormalities, syncope, cardiac conduction problems (e.g., clinically significant heart block), exercise-related cardiac events including syncope and pre syncope, or clinically significant bradycardia.
4. Subject with orthostatic hypotension or a known history of controlled or uncontrolled hypertension.
5. Subject has clinically significant ECG findings as judged by the Investigator with consideration of the central ECG laboratory's interpretation.
6. Current use of any prohibited medication or other medications, including herbal supplements, that affect BP or heart rate or that have CNS effects or affect cognitive performance, such as sedating antihistamines and decongestant sympathomimetics (inhaled bronchodilators are permitted) or a history of chronic use of sedating medications [i.e., antihistamines]) in violation of the protocol specified washout criteria at Enrolment/Visit 2.
7. Subject has used an investigational product within 30 days prior to Enrolment/Visit 2.
8. Subject is significantly overweight based on Centre for Disease Control and Prevention Body Mass Index (BMI)-for-age gender specific charts. Significantly overweight is defined as a BMI >95th percentile.
9. Children aged 6-12 years with a body weight of <25kg or adolescents aged 13-17 years with a body weight of <34kg or >91kg at Screening/Visit 1.
10. Subject has a known or suspected allergy, hypersensitivity, or clinically significant intolerance to guanfacine hydrochloride or any components found in SPD503.
11. Clinically important abnormality on drug and alcohol screen (excluding the subject's current ADHD stimulant if applicable) at Screening/Visit 1.
12. Subject has a history of alcohol or other substance abuse or dependence, as defined by DSM-IV-TR (with the exception of nicotine) within the last 6 months.
13. Subject is female and is pregnant or currently lactating.
14. Subject failed screening or was previously enrolled in this study.
15. Subject is currently considered a suicide risk in the opinion of the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation. Subjects with intermittent passive suicidal ideation are not necessarily excluded based on the assessment of the Investigator (see protocol Section 7.2.4.2 for additional guidance).
16. History of failure to respond to an adequate trial of an alpha 2-agonist for the treatment of ADHD (consisting of an appropriate dose and adequate duration of therapy in the opinion of the Investigator).
17. Subject has a history of a seizure disorder (other than a single childhood febrile seizure occurring before the age of 3 years) or the presence of a serious tic disorder (including Tourette's syndrome).
18. Subject has another member of the same household currently participating in this study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2010-05-11 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2013-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (81):
- United States (27):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - Psychiatric Centers at San Diego, Feighner Research, San Diego, California
  - Encompass Clinical Research - North Coast, Spring Valley, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Florida Clinical Research Center, LLC, Bradenton, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Amedica Research Institute, Inc., Hialeah, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - AMR-Baber Research Inc., Naperville, Illinois
  - Goldpoint Clinical Research, LLC, Indianapolis, Indiana
  - Louisiana Research Associates, Inc., New Orleans, Louisiana
  - Delmarva Family Resources, Salisbury, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Center for Psychiatry and Behavioral Medicine, Inc., Las Vegas, Nevada
  - Mount Sinai School of Medicine, New York, New York
  - Triangle Neuropsychiatry, PLLC, Durham, North Carolina
  - Ohio State University, Nisonger Center, Columbus, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc. (OCCI, Inc.), Salem, Oregon
  - CRI Worldwide, LLC, Philadelphia, Pennsylvania
  - FutureSearch Clinical Trials, Austin, Texas
  - ADHD Clinic of San Antonio, San Antonio, Texas
  - Alliance Research Group, LLC, Richmond, Virginia
  - Eastside Therapeutic Resource, Kirkland, Washington
- Belgium (8):
  - Ziekenhuis Netwerk Antwerpen, Hoboken, Antwerpen
  - Universitair Ziekenhuis Brussel, Jette, Brussels Capital
  - Universitair Ziekenhuis Gent, Ghent, Oost-vlaanderen
  - Cliniques Universitaires Saint Luc, Brussels
  - Huisartspraktijk Jaak Mortelmans, Ham
  - Centre de référence Neuropédiatrique Multidisciplinaire, Namur
  - Psypluriel, Uccle
  - Ziekenhuis Inkendaal Koninklijke Instelling v.z.w., Vlezenbeek
- Canada (4):
  - Children's and Women's Health Centre of British Columbia, Vancouver, British Columbia
  - JPM van Stralen Medicine Professional Corporation, Ottawa, Ontario
  - ADHD Clinic/The Kid's Clinic, Whitby, Ontario
  - Royal University Hospital, Saskatoon, Saskatchewan
- France (8):
  - Centre Hospitalier de Rouffach, Rouffach, Alsace
  - Hôpital Gui de Chauliac, Montpellier, Languedoc-roussillon
  - Centre Hospitalier Universitaire d'Amiens, Hôpital Nord, Amiens, Picardie
  - Hopitaux Pediatriques de Nice - CHI Lenval, Nice, Provcence Alpes Cote D'Azur
  - Centre Hospitalier Universitaire Bocage-Hôpital d'enfants, Dijon
  - Hopital Robert Debre Centre pediatrique des pathologies du sommeil, Paris
  - Hopital Robert-Debre', Paris
  - Hopital Gatien de Clocheville CHU de Tours, Tours
- Germany (9):
  - Center for Pediatric Clinical Studies, Tübingen, Baden-Wurttemberg
  - Universitätsklinik Ulm, Ulm, Baden-Wurttemberg
  - Praxis Dr. med. Dipl. Psych. Anton Lindermüller, München, Bavaria
  - Medizinisches Studienzentrum Wurzburg, Würzburg, Bavaria
  - Sozialpsychiatrisches Centrum Dr. med. Ralph Meyers, Dorsten, North Rhine-Westphalia
  - Klinikum der Johannes-Gutenberg-Universität Mainz, Mainz, Rhineland-Palatinate
  - Friedrich-Schiller-Universitat Jena, Jena, Thuringia
  - Emovis GmbH, Berlin
  - Universitatsklinikum Freiburg, Freiburg im Breisgau
- Italy (7):
  - Azienda Ospedaliera "Guido Salvini", Rho, Milan
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa
  - Azienda Ospedaliero-Universitaria Policlinico-Vittorio, Catania
  - Azienda Osp. Fatebenefratelli - Polo Territoriale UONPIA, Milan
  - Azienda ULSS 16 Padova, Padua
  - Drottning Silvias Barnsjukhus, Roma
  - Università Cattolica del Sacro Cuore, Roma
- Netherlands (3):
  - FlevoResearch, Almere Stad, Flevoland
  - Academisch Ziekenhuis Maastricht, Maastricht, Limburg
  - Mondriaan Zorggroep Heerlen, Kinder en Jeugdp sychiatrie, Maastricht
- Spain (7):
  - Hospital Son Llàtzer, Laboratorio de Neurociencias IUNICS, Palma, Balearic Islands
  - Policlínica Guipuzkoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital Fundacion Alcorcon, Alcorcón, Madrid
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Infanta Leonor, Madrid
  - Instituto Valenciano de Neurología Pediatrica, Valencia
- Barn och Ungdomsmedicin klinik Mölnlycke, Mölnlycke, Sweden
- United Kingdom (7):
  - Norfolk Community Health and Care NHS Trust, Norwich, England
  - Ryegate Children's Centre, Sheffield, England
  - Centenary House Child and Adolescent Mental Health Services, Sheffield, England
  - Queen Elizabeth II Hospital, Welwyn Garden City, England
  - Thurrock Community Hospital, Grays
  - Royal Liverpool University Hospital, Liverpool
  - Lister Hospital, Stevenage

REFERENCES:
- [Derived] Newcorn JH, Harpin V, Huss M, Lyne A, Sikirica V, Johnson M, Ramos-Quiroga JA, van Stralen J, Dutray B, Sreckovic S, Bloomfield R, Robertson B. Extended-release guanfacine hydrochloride in 6-17-year olds with ADHD: a randomised-withdrawal maintenance of efficacy study. J Child Psychol Psychiatry. 2016 Jun;57(6):717-28. doi: 10.1111/jcpp.12492. Epub 2016 Feb 12. PMID 26871297

RESULTS

PARTICIPANT FLOW:
Groups:
- Guanfacine Hydrochloride: Administered as a once-daily oral dose between 1-7mg/day depending on age and weight
- Placebo: Administered as a once-daily oral dose
Period: Open-Label Phase
Arm/Group | Guanfacine Hydrochloride | Placebo
Started | 528 | 0
Completed | 316 | 0
Not Completed | 212 | 0
Not completed — Lack of Efficacy | 56 | 0
Not completed — Response criteria not met | 46 | 0
Not completed — Adverse Event | 42 | 0
Not completed — Withdrawal by Subject | 41 | 0
Not completed — Other | 12 | 0
Not completed — Lost to Follow-up | 11 | 0
Not completed — Protocol Violation | 4 | 0
Period: Double-Blind Randomized-Withdrawal Phase
Arm/Group | Guanfacine Hydrochloride | Placebo
Started | 157 | 159
Completed | 76 | 53
Not Completed | 81 | 106
Not completed — Adverse Event | 3 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Lost to Follow-up | 3 | 2
Not completed — Lack of Efficacy | 13 | 20
Not completed — Treatment failure criteria met | 47 | 71
Not completed — Other | 4 | 3

BASELINE CHARACTERISTICS:
Population: Open-label Safety Population defined as all subjects who took at least 1 dose of any investigational product during the study. Two subjects did not receive investigational product, therefore n = 526.
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 526
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.7 (2.7)
Age, Customized [Count of Participants; unit: Participants]
  6-12 years | 391
  13-17 years | 135
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130
  Male | 396
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 19
  CANADA | 30
  FRANCE | 14
  GERMANY | 27
  ITALY | 31
  NETHERLANDS | 29
  SPAIN | 68
  SWEDEN | 5
  UNITED KINGDOM | 25
  UNITED STATES | 278

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Failures During the Double-Blind Randomized-Withdrawal Phase
Description: Treatment failure was defined as >= 50% increase (worsening) in ADHD-RS-IV total score and a >= 2 point increase (worsening) in CGI-S score compared with the respective scores at the Double-blind Randomized-withdrawal Baseline Visit at 2 consecutive Double-blind Randomized-withdrawal Phase visits. Subjects meeting these criteria were regarded as treatment failures regardless of whether or not they were withdrawn. All subjects who discontinued the study for any reason were regarded as treatment failures for the primary analysis.
Time Frame: 26 weeks
Population: Randomized Full Analysis Set (FAS) defined as all subjects who were randomized and took at least 1 dose of investigational product during the Double-blind Randomized-withdrawal Phase. Subjects from Site 801 were excluded from the Randomized FAS.
Measure: Number (95% Confidence Interval); unit: percentage of treatment failures
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 151 | 150
percentage of treatment failures | 64.9 [57.3 to 72.5] | 49.3 [41.3 to 57.3]
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.006, Cochran-Mantel-Haenszel; Difference in treatment failures = -15.6, 95% CI 2-sided [-26.6 to -4.5]

2. Secondary Outcome: Time to Treatment Failure During the Double-Blind Randomized-Withdrawal Phase
Description: as for outcome 1
Time Frame: 26 weeks
Population: Randomized FAS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 151 | 150
Days | 56.0 [44.0 to 97.0] | 218.0 [118.0 to NA] — There were not enough treatment failure events by study completion to calculate an upper CI.
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.003, Log Rank

3. Secondary Outcome: Change From Double-Blind Randomized-Withdrawal Baseline in Attention Deficit Hyperactivity Disorder Rating Scale-fourth Edition (ADHD-RS-IV) Total Score at Week 26 of the Double-Blind Randomized-Withdrawal Phase - Last Observation Carried Forward (LOCF)
Description: The ADHD-RS-IV consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and week 26
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 151 | 150
units on a scale | 15.89 (1.225) | 9.64 (1.21)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -6.24, 95% CI 2-sided [-9.01 to -3.48]

4. Secondary Outcome: Percent of Subjects With an Assessment of Normal/Borderline Mentally Ill on Clinical Global Impression-Severity of Illness (CGI-S) Scale During the Double-Blind Randomized-Withdrawal Phase - LOCF
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale: 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill)
Time Frame: 26 weeks
Population: Randomized FAS
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 151 | 150
percentage of subjects | 32.5 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.001, Cochran-Mantel-Haenszel — Nominal p-value uncorrected for multiplicity; Difference in percent of subjects = 17.5, 95% CI 2-sided [6.6 to 28.5]

5. Secondary Outcome: Change From Double-Blind Randomized-Withdrawal Baseline in the Weiss Functional Impairment Rating Scale - Parent Report (WFIRS-P) Global Score at Week 26 of the Double-Blind Randomized-Withdrawal Phase - LOCF
Description: The WFIRS-P is a 50-item scale with each item scored from 0 (never/not at all) to 3 (very often/very much). Mean scores range from 0 to 3. Higher scores indicate greater functional impairment.
Time Frame: Baseline and week 26
Population: Randomized FAS
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 151 | 150
units on a scale | 0.23 (0.036) | 0.16 (0.035)
Statistical Analysis 1: Comparison: Placebo vs Guanfacine Hydrochloride; Test type: Superiority or Other; p = 0.118, ANCOVA — Nominal p-value uncorrected for multiplicity; Difference in Least Squares Mean = -0.06, 95% CI 2-sided [-0.14 to 0.02]

6. Secondary Outcome: Health Utilities Index-2/3 (HUI 2/3) Scores During the Double-Blind Randomized-Withdrawal Phase - LOCF
Description: HUI is used to describe health status and to obtain utility scores by collecting data using one or more questionnaires in formats selected to match the specific study design criteria. Scoring ranges from 0.00 (dead) to 1.00 (perfect health). Higher scores represent better health status.
Time Frame: 26 weeks
Population: Randomized FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 142 | 138
units on a scale | 0.899 (0.1272) | 0.900 (0.1229)

7. Secondary Outcome: Columbia-Suicide Severity Rating Scale During Double-Blind Randomized-Withdrawal Phase
Description: C-SSRS is a semi-structured interview that captures the occurence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The interview includes definitions and suggested questions to solicit the type of information needed to determine if a suicide-related thought or behaviour occurred. The assessment is done by the nature of the responses, not by a numbered scale.
Time Frame: 26 weeks
Population: Randomized Safety Population defined as all subjects who were randomized and who took at least 1 dose of investigational product during the Double-blind Randomized-withdrawal Phase.
Measure: Number; unit: participants
Arm/Group | Placebo | Guanfacine Hydrochloride
Number analyzed (Participants) | 158 | 157
participants
  Suicidal ideation | 2 | 2
  Suicidal behavior | 0 | 0

8. Secondary Outcome: Change From Open-Label Baseline in ADHD-RS-IV Total Score at Week 13 of the Open-Label Phase - LOCF
Description: as for outcome 3
Time Frame: Baseline and 13 weeks
Population: Open-label Full Analysis Set (FAS) defined as all subjects who took at least 1 dose of any investigational product during the study. The Subjects from Site 801 were excluded from the Open-label FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 497
units on a scale | -25.2 (11.97)
Statistical Analysis 1: Comparison: Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Nominal p-value uncorrected for multiplicity

9. Secondary Outcome: Percentage of Responders in the Open-Label Phase - LOCF
Description: Response is defined as a percentage decrease (improvement) from Baseline in the ADHD-RS-IV total score of >=30% and a CGI-S score of 1 or 2.
Time Frame: 13 weeks
Population: Open-label FAS
Measure: Number; unit: percentage of participants
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 497
percentage of participants | 68.6

10. Secondary Outcome: Percent of Subjects With Improvement on Clinical Global Impression-Improvement (CGI-I) Scores During Open-Label Phase - LOCF
Description: Clinical Global Impression-Improvement (CGI-I) consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 13 weeks
Population: Open-label FAS
Measure: Number; unit: percentage of participants
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 497
percentage of participants | 76.1

11. Secondary Outcome: Percent of Subjects With an Assessment of Normal/Borderline Mentally Ill on CGI-S Scale During the Open-Label Phase - LOCF
Description: as for outcome 4
Time Frame: 13 weeks
Population: Open-label FAS
Measure: Number; unit: percentage of participants
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 503
percentage of participants | 68.9

12. Secondary Outcome: Change From Open-Label Baseline in WFIRS-P Global Score at Week 13 of the Open-Label Phase - LOCF
Description: as for outcome 5
Time Frame: Baseline and week 13
Population: Open-label FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 405
units on a scale | -0.35 (0.414)
Statistical Analysis 1: Comparison: Guanfacine Hydrochloride; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Nominal p-value uncorrected for multiplicity

13. Secondary Outcome: HUI 2/3 Scores During the Open-Label Phase - LOCF
Description: as for outcome 6
Time Frame: 13 weeks
Population: Open-label FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 417
units on a scale | 0.892 (0.1230)

14. Secondary Outcome: Columbia-Suicide Severity Rating Scale During Open-Label Phase
Description: as for outcome 7
Time Frame: 13 weeks
Population: Open-label Safety Population defined as all subjects who took at least 1 dose of any investigational product during the study.
Measure: Number; unit: participants
Arm/Group | Guanfacine Hydrochloride
Number analyzed (Participants) | 526
participants
  Suicidal ideation | 1
  Suicidal behavior | 2

ADVERSE EVENTS:
Description: Open-label and Randomized Safety Populations consist of all subjects who took at least 1 dose of investigational product during their specific Phase. Two subjects in the Open-label Phase (n=526) and one subject in the Randomized-withdrawal Phase (n=315) did not receive investigational product and were excluded from their respective populations.
Groups:
- Guanfacine Hydrochloride (Open-Label Phase); Guanfacine Hydrochloride (Randomized-Withdrawal Phase): Administered as a once-daily oral dose between 1-7mg/day depending on age and weight
- Placebo (Randomized-Withdrawal Phase): Administered as a once-daily oral dose
Arm/Group | Guanfacine Hydrochloride (Open-Label Phase) | Placebo (Randomized-Withdrawal Phase) | Guanfacine Hydrochloride (Randomized-Withdrawal Phase)
Serious Adverse Events (participants affected / at risk) | 5/526 | 4/158 | 2/157
Other Adverse Events (participants affected / at risk) | 423/526 | 51/158 | 65/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine Hydrochloride (Open-Label Phase) (N=526) | Placebo (Randomized-Withdrawal Phase) (N=158) | Guanfacine Hydrochloride (Randomized-Withdrawal Phase) (N=157)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Conduct disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Family stress (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Guanfacine Hydrochloride (Open-Label Phase) (N=526) | Placebo (Randomized-Withdrawal Phase) (N=158) | Guanfacine Hydrochloride (Randomized-Withdrawal Phase) (N=157)
Abdominal pain upper (Gastrointestinal disorders) | 60 (70) | 8 (10) | 3 (4)
Constipation (Gastrointestinal disorders) | 31 (38) | 3 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 37 (46) | 3 (4) | 4 (5)
Nausea (Gastrointestinal disorders) | 33 (42) | 4 (4) | 5 (5)
Fatigue (General disorders) | 130 (186) | 2 (2) | 8 (11)
Irritability (General disorders) | 37 (41) | 3 (3) | 2 (2)
Nasopharyngitis (Infections and infestations) | 36 (39) | 13 (14) | 11 (14)
Upper respiratory tract infection (Infections and infestations) | 31 (33) | 10 (10) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 30 (32) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 50 (62) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 144 (242) | 18 (24) | 25 (34)
Sedation (Nervous system disorders) | 47 (61) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 254 (386) | 0 (0) | 19 (27)
Hypotension (Vascular disorders) | 29 (32) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 9 (11) | 5 (6)
Pyrexia (General disorders) | 22 (28) | 5 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.